CLINICAL TRIAL: NCT06312293
Title: Transcutaneous Auricular Vagus Nerve Stimulation: Comparison of Effectiveness of In-ear and Behınd-ear Stimulation
Brief Title: Comparison of Effectiveness In-ear and Behind-ear Vagus Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Principal Investigator, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: STUDYAP0004
Record Dates: First submitted 2024-01-03; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- In-Ear stimulation (Experimental): Participants in this group underwent intra-ear transcutaneous vagus nerve simulation.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- Behind the ear stimulation (Experimental): Participants in this group underwent transcutaneous vagus nerve simulation behind the ear.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- In-Ear stimulation (device switched off) (Placebo Comparator): In order to see the placebo effect of in-ear simulation in participants in this group, the electrode was placed inside the ear with the device closed and the results were evaluated.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation
- Behind the ear stimulation (device switched off) (Placebo Comparator): In order to see the placebo effect of behind-ear simulation in participants in this group, the electrode was placed inside the ear with the device closed and the results were evaluated.
  Interventions: Device: Transcutaneous Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Vagus Nerve Stimulation — All techniques used to stimulate the vagal nerve are called vagus nerve stimulation.

SUMMARY:
The use of vagus nerve stimulation (VSS), one of the examples of neuromodulation therapies, continues to increase in the medical field. Basically, invasive (iVSS) and transcutaneous VSS (tVSS) can be performed. tVSS is more preferred because of its advantages such as easy application, not requiring surgical procedure and having fewer side effects. VSS has long been an approved treatment modality in the treatment of epilepsy and refractory depression. tVSS can be administered from the auricular-auricular or posterior ear region. The vagus nerve (VS) belongs to the parasympathetic branch of the autonomic nervous system and has an effect on vital functions. There are also studies in the literature showing that VS stimulation reduces inflammation. In addition to this effect, the vagus nerve may also show analgesic activity through pain-related pathways. Due to its anti-inflammatory and analgesic effects, VSS has become a new treatment method in diseases in which various inflammatory processes are shown in the etiology such as inflammatory bowel diseases, musculoskeletal system diseases and central nervous system diseases.

DETAILED DESCRIPTION:
There are no generally accepted values for taVNS (transcutaneous auricular vagus nerve stimulation) application parameters (amplitude, frequency, intensity, duration, side); therefore, there are heterogeneous applications in studies. In a meta-analysis on the safety profile of taVSS, local skin irritation (18. 2%), headache (3.6%), nasopharyngitis (1.7%), dizziness (1.4%) and nausea (1.1%) were reported and taVSS treatment was reported as an effective and safe treatment with these side effects, most of which were transient and did not require additional intervention.

During taVNS, autonomic activities increase in favour of the parasympathetic system and this results in an increase in heart rate variability (HRV). Although an increase in HRV has been demonstrated by different studies, the factors that can predict the change in HRV are not clear. In a study by Geng et al. using taVSS, it was observed that HRV indicators representing vagal nerve activity increased significantly when stimulation was performed in the morning, but evening stimulation did not yield similar results. In addition, they found that improvements in measures of autonomic balance were more pronounced in the presence of lower vagal activity; they also found that by increasing the duration of stimulation, the effect of taVNS on HRV was not regulated by duration. In other words, HRV changes had the best effect only at the beginning of stimulation.

ELIGIBILITY:
Inclusion Criteria:

* To be 18 years of age or older,
* Not having any acute or chronic health problems,
* No previous transcutaneous vagus nerve stimulation application.

Exclusion Criteria:

* Using drugs, alcohol or smoking
* Being in the post menopausal phase
* Pregnancy history
* Known history of acute or chronic illness
* Having received any medication affecting the autonomic nervous system

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | Baseline and immediately after the intervention
  The effectiveness of vagus nerve stimulation, its effect on autonomic nervous system activity was evaluated using heart rate variability. Polar H7 device was used for this. The heart rate was recorded non-invasively over the chest for 5 minutes and the beat-to-beat (R-R) variability was measured with Kubios software.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Erenler, Prof. Dr., Study Chair — Igdir University
Locations (1):
- Igdir University, Iğdır, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Szeles JC, Kampusch S, Thurk F, Clodi C, Thomas N, Fichtenbauer S, Schwanzer C, Schwarzenberger S, Neumayer C, Kaniusas E. Bursted auricular vagus nerve stimulation alters heart rate variability in healthy subjects. Physiol Meas. 2021 Oct 29;42(10). doi: 10.1088/1361-6579/ac24e6. PMID 34496357
- [Background] Clancy JA, Mary DA, Witte KK, Greenwood JP, Deuchars SA, Deuchars J. Non-invasive vagus nerve stimulation in healthy humans reduces sympathetic nerve activity. Brain Stimul. 2014 Nov-Dec;7(6):871-7. doi: 10.1016/j.brs.2014.07.031. Epub 2014 Jul 16. PMID 25164906
- [Background] Carandina A, Rodrigues GD, Di Francesco P, Filtz A, Bellocchi C, Furlan L, Carugo S, Montano N, Tobaldini E. Effects of transcutaneous auricular vagus nerve stimulation on cardiovascular autonomic control in health and disease. Auton Neurosci. 2021 Dec;236:102893. doi: 10.1016/j.autneu.2021.102893. Epub 2021 Oct 9. PMID 34649119
- [Background] Trevizol AP, Shiozawa P, Taiar I, Soares A, Gomes JS, Barros MD, Liquidato BM, Cordeiro Q. Transcutaneous Vagus Nerve Stimulation (taVNS) for Major Depressive Disorder: An Open Label Proof-of-Concept Trial. Brain Stimul. 2016 May-Jun;9(3):453-454. doi: 10.1016/j.brs.2016.02.001. Epub 2016 Feb 10. No abstract available. PMID 26944188
- [Background] Peng X, Baker-Vogel B, Sarhan M, Short EB, Zhu W, Liu H, Kautz S, Badran BW. Left or right ear? A neuroimaging study using combined taVNS/fMRI to understand the interaction between ear stimulation target and lesion location in chronic stroke. Brain Stimul. 2023 Jul-Aug;16(4):1144-1153. doi: 10.1016/j.brs.2023.07.050. Epub 2023 Jul 28. PMID 37517466